CLINICAL TRIAL: NCT06965010
Title: Hybrid Clinical Effectiveness Trial Type II of Measurement Based Care in Opioid Treatment Programs
Brief Title: Measurement Based Care in Opioid Treatment Programs
Status: Enrolling by invitation | Phase: Not Applicable | Type: Interventional
Sponsor: University of Pittsburgh (Other)
Collaborators: National Institute on Drug Abuse (NIDA) (NIH)
Responsible Party: Principal Investigator, Renee Cloutier, Assistant Professor of Medicine, University of Pittsburgh
Allocation: Randomized | Model: Sequential | Masking: None | Purpose: Treatment
Other Study IDs: STUDY24080133; 1RM1DA059395-01 (NIH)
Record Dates: First submitted 2025-04-09; First posted 2025-05-11 (Actual); Last update posted 2025-11-10 (Actual); Status verified 2025-11

CONDITIONS: Opioid Use Disorder
MeSH Terms: conditions — Opioid-Related Disorders | interventions — Weights and Measures

STUDY DESIGN:
Intervention Model Description: This study is a hybrid implementation effectiveness type II trial with a stepped wedge design. Each cohort of OTP sites (~5 sites per cohort; 4 cohorts or 20 OTP sites total) will begin in the Measurement as Usual condition (MAU) and then cross over to a 9-month MBC+ Implementation Phase followed by a Sustainability Phase to monitor ongoing MBC implementation. Individual participant may experience one or the other or both interventions
Oversight: Data Monitoring Committee: Yes | FDA-regulated Drug: No | FDA-regulated Device: No

ARMS (3):
- Measurement Based Care (Experimental): Monthly Use of Measurement-Based Care using Greenspace Mental Health tools
  Interventions: Behavioral: Measurement-based care
- Measurement As Usual followed by Measurement Based Care (Experimental): Participation in existing processes available within treatment sites including semi structured interviews followed by monthly use of Measurement-Based Care using Greenspace Mental Health tools
  Interventions: Behavioral: Measurement-based care; Behavioral: Measurement As Usual
- Measurement As Usual (Active Comparator): Participation in existing processes available within treatment sites including semi structured interviews
  Interventions: Behavioral: Measurement As Usual

INTERVENTIONS:
Behavioral: Measurement-based care — Patients will complete MBC measures with their treatment provider and follow-up surveys conducted at baseline and monthly intervals. Both providers and patients will use the Greenspace Mental Health tools to regularly assess patient-reported symptoms, review results together, and collaboratively design individualized treatment plans. Providers will implement MBC to guide treatment adjustments based on these assessments.
  Arms: Measurement As Usual followed by Measurement Based Care; Measurement Based Care
Behavioral: Measurement As Usual — Patients will participate in Measurement As Usual (MAU) via the existing processes available within treatment sites. Currently, patients are assessed and participate in semi-structured interviews at 6-month increments to assess progress and appropriateness of level of care.
  Arms: Measurement As Usual; Measurement As Usual followed by Measurement Based Care

SUMMARY:
The goal of this HEAL Initiative study is to enhance the measurement, quality, and equity of care delivered in 20 community opioid treatment programs (OTPs) by creating and using measurement-based care (MBC) tools and systems. Patients will use MBC tools to track their symptoms and discuss with their providers. This data will be collected over the course of the study to evaluate the effectiveness of MBC in improving patient care and treatment outcomes.

DETAILED DESCRIPTION:
Opioid use disorder (OUD) remains a critical public health crisis in Pennsylvania. Measurement-based care (MBC) is the systematic use of client self-report data to inform treatment and is an evidence-based intervention that is uniquely well suited to complement opioid use disorder (OUD) pharmacotherapy that occurs within opioid treatment programs (OTPs). The study aims to enhance the measurement, quality, and equity of care delivered in 20 community OTPs by co-designing and implementing MBC tools and systems. Using a Hybrid Implementation Effectiveness Type II trial with a stepped-wedge design, MBC implementation (e.g., fidelity) and clinical (e.g., patient retention, improved quality of life) effectiveness will be evaluated simultaneously with quantitative and qualitative data. This study aims to provide: (1) preliminary evidence regarding the role and significance of capitalizing on MBC in opioid use disorder (OUD) treatments (including evidence on potential mechanisms underlying MBC's effects); (2) enhanced adoption of MBC via implementation strategies that are co-designed with stakeholders (policymaker, payer, and OTP); and (3) alternative avenues to potentially enhance symptom-related outcomes and treatment retention of OUD interventions with downstream societal, psychological, and public health benefits.

ELIGIBILITY:
Inclusion Criteria

OTP patients will be eligible to participate if they:

1. are adults (aged 18 years or older);
2. are initiating MOUD at the OTP, as a new patient (as defined by OTP guidelines); and
3. speak primarily English or Spanish.

Exclusion Criteria

OTP patients will be excluded from participation if they:

1. are under the age of 18;
2. are not a new MOUD patient at the OTP
3. do not speak primarily English or Spanish.

Min Age: 18 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Enrollment: 3650 (Estimated)
Dates: Start 2025-10-01 (Actual); Primary Completion 2027-11-01 (Estimated); Study Completion 2028-08-31 (Estimated)

PRIMARY OUTCOMES:
Change in Patient Treatment Retention - Clinical Effectiveness Outcome | Continuous following new MOUD patient intake events during the 9-month periods prior to and during MBC+/Implementation Phase in an OTP
  Change in Patient Treatment Retention: clinic-level outcome measure that tracks the duration of OUD treatment based on medications, counseling and related services, as recorded in the claims data. Specific measures are the (1) % of patients still in treatment 6 months after initiating MOUD and (2) the average number of months new MOUD patients remain in treatment (12-month follow-up window).
Change in Patient's Perceived Recovery - Clinical Effectiveness Outcome | Monthly during the 9-month MBC+/Implementation Phase, sub-group of OTP sites during 9-month period pre-MBC+/Implementation Phase
  Change in Patient Recovery: patient-level outcome measure that evaluates progress in patient recovery obtained from survey data. The Brief Addiction Monitoring assessment question will be administered monthly to monitor substance use.
Change in Patient Quality of Life - Clinical Effectiveness Outcome | At baseline and every 3 months during the 9-month MBC+/Implementation Phase, sub-group of OTP sites during 9-month period pre-MBC+/Implementation Phase
  Change in Patient Quality of Life: patient-level outcome measure that evaluates progress in patient quality of life. The Patient-Reported Outcomes Measurement Information System (PROMIS-29) Instrument will be administered at baseline and at every 3 months to evaluate and monitor physical, mental, and social health via The Greenspace Mental Health tool.
Sustainment of Measurement-Based Care Implementation | During the Sustainment Phase ~9 months post-Implementation
  The sustainment of MBC implementation is defined as the extent to which providers continue to use MBC tools with fidelity following the removal of active implementation support, based on data sourced from Greenspace and/or provider surveys. Each treatment session will continue to receive a score of "1" for documentation of MBC data collection, a "2" for documented data sharing, and a "3" for documented action informed by data. Sessions without MBC documentation will receive a "0." Sustainability is assessed by examining whether fidelity to core MBC components is maintained over time. Potential metrics include:
  Percentage of sessions with completed MBC assessments during Sustainment Percentage of sessions where MBC results were reviewed with patients during Sustainment Percentage of sessions with documented action taken during Sustainment Percentage of providers meeting a predefined threshold for sustained fidelity (e.g., 80% of sessions scoring ≥2) during Sustainment
Fidelity of Measurement-Based Care Implementation | Monthly during the 9-month MBC+/Implementation Phase
  The Fidelity of MBC Implementation is defined as the extent to which providers administer and use MBC tools as intended based on data sourced from Greenspace and/or provider surveys during the Implementation Phase. MBC fidelity will be a single outcome measure that ranges from 0-3. Each treatment session will receive a "1" for documentation of MBC data collection, a "2" for documented data sharing, and a "3" for documented action informed by data. All attended appointments without MBC documentation will receive a "0."
  Potential metrics include:
  Percentage of sessions with completed MBC assessments Percentage of sessions where MBC results were reviewed with patients Percentage of sessions with documented action taken
Adoption of Measurement-Based Care Implementation as Assessed by Patient Surveys - Measure Implementation Outcome | Monthly during the 9-month MBC+/Implementation Phase
  The adoption of MBC implementation will be assessed based on the percentage of OTP treatment providers who use MBC during and after active implementation. Adoption will be measured using patient surveys during the Implementation Phase.
Adoption of Measurement-Based Care Implementation as Assessed by Greenspace Mental Health tools - Measure Implementation Outcome | Monthly during the 9-month MBC+/Implementation Phase
  The adoption of MBC implementation will be assessed based on the percentage of OTP treatment providers who use MBC during and after active implementation. Adoption will be measured using Greenspace Mental Health tools during the Implementation Phase.

OTHER OUTCOMES:
Net costs to Medicaid and cost-effectiveness | From the beginning of 36 Month stepped wedge trial timeline and 9-month MBC+/Implementation Phase through the completion of the 6-month Sustainability Phase
  A health economic analysis will calculate net costs to Medicaid of all-cause healthcare use by the patients. These costs will be based on each patient's healthcare claims for Medicaid reimbursement. Each service unit recorded in the claims data will be converted to its 2028 $US value and summed to create a total cost in $. In addition to costs from Medicaid patient claims, we will estimate the programmatic costs in the MBC+/Implementation Phase using activity-based costing which collects resource data (staff labor, space, materials, equipment, and software) and unit costs (wages, prices, subcontract amounts) needed to implement MBC+. Using the net Medicaid costs and Patient Treatment Retention outcome, we will estimate the cost-effectiveness of MBC+. Cost-effectiveness is the ratio of the difference in costs to the difference in outcome between the MBC+ sample and the MAU sample. In this case, that is the cost to Medicaid needed to improve treatment retention rates by 1 add'l % point.

CONTACTS AND LOCATIONS:
Overall Officials: Renee Cloutier, PhD, Principal Investigator — University of Pittsburgh; Kelli S Scott, PhD, Principal Investigator — Northwestern University Feinberg School of Medicine; Arnie Aldridge, PhD, Principal Investigator — RTI International
Locations (1):
- The University of Pittsburgh, Pittsburgh, Pennsylvania, United States

IPD SHARING:
Plan to Share IPD: Yes
Identifiable data will not be shared from this research project. HEAL-MBC will work with NIDA to develop a plan consistent with the HEAL Initiative Public Access and Data Sharing Policy to ensure that Harm Reduction Network Publications and, to the extent possible, the underlying primary data are immediately and broadly available to the public in a way that protects participant data in accordance with 45 C.F.R. 46 and other applicable laws. The data sharing plan will comply with the Health Insurance Portability and Accountability Act (HIPAA) of 1996 regulations and Institutional Review Board requirements. Data will be submitted to the NIDA-supported National Addiction & HIV Data Archive Program (NAHDAP) repository for storage, archiving, and sharing for future studies.
Time Frame: Raw data will be deposited to NAHDAP throughout the study as it is received. Cleaned analytic data files will be deposited to NAHDAP within 12 months of receiving the final assessment for the final participant.
Access Criteria: Authorized research personnel who are trained in the ethical conduct of research (e.g., Collaborative Institutional Training Initiative, National Institutes of Health tutorials) will have access to the research laboratory and participant data.